CLINICAL TRIAL: NCT04035460
Title: A Pilot Randomized Controlled Study of Non-invasive Oxygenation and Ventilation in Patients With Acute Hypoxemic Respiratory Failure (AHRF): A Comparison of Oxygen Delivery Via Helmet Interface Versus High Flow Nasal Cannula (HFNC)
Brief Title: A Pilot Study Comparing Oxygen Delivery Via Helmet Interface Versus High Flow Nasal Cannula
Acronym: NOVA-pilot
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Baystate Medical Center (Other)
Responsible Party: Principal Investigator, Mark Tidswell, Associate Professor of Medicine and Surgery, Baystate Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 952633
Record Dates: First submitted 2019-07-16; First posted 2019-07-29 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Hypoxemic Respiratory Failure
Keywords: non-invasive ventilation
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Head Protective Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Helmet oxygenation group (Active Comparator): Patients randomized to helmet NIPPV will receive noninvasive oxygenation and ventilation via a latex free helmet
  Interventions: Device: Helmet
- High Flow Nasal Oxygen (Active Comparator): Oxygen will be passed through a heated humidifier and applied continuously through large-bore nasal prongs
  Interventions: Device: High Flow Nasal Oxygen

INTERVENTIONS:
Device: Helmet — The helmet encloses the head and neck of the patient, has a rigid ring and is secured by 2 armpit braces. A soft collar adheres to the neck and ensures a sealed connection once the helmet is inflated.
  Arms: Helmet oxygenation group
Device: High Flow Nasal Oxygen — Large-bore nasal prongs through which oxygen is delivered at high flow rates
  Arms: High Flow Nasal Oxygen

SUMMARY:
Our main objective is to collect feasibility data on helmet NIPPV and other clinical elements in to eventually prepare for a full scale randomized trial based on findings of this pilot study.

DETAILED DESCRIPTION:
Patients with acute hypoxemia leading to respiratory failure are frequently supported by endotracheal intubation and mechanical ventilation. Unfortunately an invasive approach to support is associated with risks of lung injury, infection, need for heavy sedation, and increased mortality. Non-invasive oxygen delivery, by mask (BiPAP or CPAP), high flow nasal cannula or helmet interface, is better tolerated and reduces risks associated with invasive mechanical ventilation. A growing body of medical literature and clinical experience suggests that non-invasive oxygen delivery can prevent the need for endotracheal intubation in some patients. This proposal will compare two different modes of non-invasive oxygen delivery: helmet and high flow nasal cannula.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. AHRF defined as:

   A ratio of partial pressure of oxygen (PaO2) to fraction of inspired oxygen (FiO2) between 100 - 250 mm Hg while breathing O2 from Venturi mask, or other delivery system that allows quantification of FiO2 such as Mask-NIPPV or HFNC.

   When no arterial blood gas (ABG) result available, use transcutaneous oxygen saturation measurement (SpO2) to impute PaO2 (Appendix A.2 for Table of PaO2 / FiO2 imputed from SpO2 [Brown 2017]. If no oxygenation data prior to use of Mask-NIPPV or HFNC are available, then P/F ratio 100 - 250 on Mask-NIPPV or HFNC meets this criterion.
3. Respiratory rate (RR) ≥24 /min and/or subjective shortness of breath (Modified Borg Dyspnea Scale ≥ 2)

Exclusion Criteria:

1. P/F Ratio < 100 (Severe ARDS) on quantifiable FiO2
2. More than 24 hours has elapsed since the patient met criteria for AHRF (Inclusion #2 and 3, above)
3. Urgent need for intubation

   Criteria for intubation:

   i. RR>40 ii. Lack of improvement of respiratory muscle fatigue iii. Copious tracheal secretions that require frequent suctioning iv. Acidosis with a potential Hydrogen (pH) <7.35 v. Acute hypercarbia (PaCO2 > 45 mm Hg) vi. SpO2 < 88% for more than 5 minutes despite FiO2 and non-invasive support vii. Respiratory or cardiac arrest viii. Glasgow Coma Scale ≤ 8
4. Contraindication to HFNC, Helmet-NIPPV, or Mask-NIPPV
5. Upper airway obstruction, facial trauma
6. Copious secretions, airway bleeding, epistaxis or vomiting
7. Primary cause of respiratory failure is exacerbation of chronic obstructive pulmonary disease (COPD) or asthma
8. Elevated intracranial pressure >20 mm Hg
9. Home mechanical ventilation except for CPAP/BiPAP used solely for sleep disordered breathing
10. Persistent hemodynamic instability (systolic blood pressure (SBP)<90 or mean arterial pressure (MAP)<60 despite IV fluid resuscitation, or norepinephrine dose > 0.1 mcg/kg/min or equivalent vasopressor dose)
11. Plan for procedure during which NIPPV or HFNC is contraindicated. Okay to enroll if procedure is complete and AHRF persists within 24 hours.
12. Absence of airway protective gag reflex or cough
13. Tracheostomy
14. Lack of informed consent
15. Pregnancy
16. Actual body weight exceeding 1 kg per cm of height
17. Diffuse alveolar hemorrhage
18. Severe acute pancreatitis as etiology for hypoxemia
19. Recent upper gastrointestinal surgical anastomosis within the past 30 days
20. Enrollment in another clinical trial within the past 30 days
21. Unsuitable for non-invasive ventilation in the judgment of the treating MD
22. Decision to withhold life-sustaining treatment. Patients with Do-Not-Resuscitate (DNR) or No Cardiopulmonary resuscitation (No CPR) order may be enrolled.
23. Do not intubate order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Rate of intubation | 28 days
  To determine the rates of intubation for subjects with Acute Hypoxemic Respiratory Failure (AHRF) managed by non-invasive modalities High Flow Nasal Cannula (HFNC) and Helmet NIPPV.

SECONDARY OUTCOMES:
Time to intubation | 28 days
  Hours and minutes from time of initiation of protocol until intubation
Intubation-free days through day 28 | 28 days
  number of days from the time of randomization to day 28 after randomization on which the patient is not intubated and does not require invasive mechanical ventilation
Organ-failure-free days through day 28 | 28 days
  Daily determination of presence or absence of Cardiovascular, Kidney, Liver, Central Nervous System, and Hematological Dysfunction.
Mortality prior to discharge from hospital (up to study day 90 whichever comes first) | 90 days
  hospital mortality
Hospital mortality to day 28 | 28 days
  hospital mortality
ICU free-days to day 28 | 28 days
  days not in ICU
Hospital length of stay | 28 days
  duration of hospital stay
Rate of cross-over between groups | 28 days
  The percentage of patients in each group crossed over to the alternative group or another form of noninvasive ventilation.
Complications | 28 days
  Adverse events other than failure of the noninvasive oxygenation device
Ventilator associated pneumonia, barotrauma | 28 days
  Complications due to mechanical ventilation
Total daily dose of sedative medications (milligram) | 7 days
  Assessment of Sedation medications
Highest level of daily mobility through day 7 | 7 days
  Activity level
Tolerance of the devices | 28 days
  Daily assessment with visual analog scale for comfort, range 0-5, with 0= no discomfort and 5=unable to tolerate
Rate and reason for exclusion from enrollment to this trial of Helmet-NIPPV vs. HFNC | through study completion, an average of 1 year
  Reasons for exclusion of patients meeting inclusion criteria
Rate of intubation in non-enrolled patients that meet inclusion and exclusion criteria | 28 days
  Usual care comparison
Richmond Agitation and Sedation Scale (RASS) | 7 days
  Highest daily RASS score. The scale range is -5 to +4 in integer increments, Where -5 is unarousable, 0 is alert and calm, and +4 is combative
Confusion Assessment Method for the ICU (CAM-ICU) | 7 days
  Daily assessment of presence or absence of delirium

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Tidswell, MD, Principal Investigator — Baystate Medical Center
Locations (1):
- Baystate Medical Center, Springfield, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No